CLINICAL TRIAL: NCT05204381
Title: Causal Role of Theta and Alpha Oscillations in Output-gating
Brief Title: Theta Connectivity in Working Memory
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-0248; 1R01MH124387 (NIH)
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-01

CONDITIONS: Executive Function

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Theta Stimulation (Experimental): Rhythmic transcranial magnetic stimulation (TMS) is delivered to frontal and parietal cortex during performance of a cognitive control task while electroencephalography (EEG) is recorded. In the fourth and fifth sessions, stimulation is delivered in near-zero phase lag theta-frequency, anti-synchrony theta-frequency, near-zero phase lag arrhythmic-in-synchrony stimulation, and arrhythmic-independent stimulation. The near-zero phase lag arrhythmic-in-synchrony stimulation and arrhythmic-independent stimulation is delivered in both the fourth and fifth session to serve as an active control. Each session is separated by at least one day as a washout period.
  Interventions: Device: Theta-frequency near-zero phase lag stimulation; Device: Theta-frequency anti-synchrony stimulation; Device: Arrhythmic near-zero phase lag stimulation; Device: Arrhythmic independent stimulation
- Alpha Stimulation (Experimental): Rhythmic transcranial magnetic stimulation (TMS) is delivered to frontal and parietal cortex during performance of a cognitive control task while electroencephalography (EEG) is recorded. In the fourth and fifth sessions, stimulation is delivered in near-zero phase lag alpha-frequency, anti-synchrony alpha-frequency, near-zero phase lag arrhythmic-in-synchrony stimulation, and arrhythmic-independent stimulation. The near-zero phase lag arrhythmic-in-synchrony stimulation and arrhythmic-independent stimulation is delivered in both the fourth and fifth session to serve as an active control. Each session is separated by at least one day as a washout period.
  Interventions: Device: Arrhythmic near-zero phase lag stimulation; Device: Arrhythmic independent stimulation; Device: Alpha-frequency near-zero phase lag stimulation; Device: Alpha-frequency anti-synchrony stimulation

INTERVENTIONS:
Device: Theta-frequency near-zero phase lag stimulation — Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in theta-frequency (approximately 6 Hz) with a near-zero phase lag.
  Arms: Theta Stimulation
Device: Theta-frequency anti-synchrony stimulation — Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in theta-frequency (approximately 6 Hz) with a 180 degree phase offset, anti-synchrony.
  Arms: Theta Stimulation
Device: Arrhythmic near-zero phase lag stimulation — Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in an arrhythmic pattern with a near-zero phase lag matched in duration to the rhythmic stimulation for that session.
Device: Arrhythmic independent stimulation — Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in different independent arrhythmic patterns matched in duration to the rhythmic stimulation for that session.
Device: Alpha-frequency near-zero phase lag stimulation — Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in alpha-frequency (approximately 10 Hz) with a near-zero phase lag.
  Arms: Alpha Stimulation
Device: Alpha-frequency anti-synchrony stimulation — Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in alpha-frequency (approximately 10 Hz) with a 180 degree phase offset, anti-synchrony.
  Arms: Alpha Stimulation

SUMMARY:
The participants will perform a cognitive control task. During the task, rhythmic trains of transcranial magnetic stimulation will be delivered to the prefrontal cortex and parietal cortex. Participants will be screened for their ability to perform the task. Magnetic resonance imaging will be used to localize regions of interest to be targeted. Electroencephalography will be collected concurrent with stimulation.

DETAILED DESCRIPTION:
This study is a pilot, five-session study with transcranial magnetic stimulation (TMS), electroencephalography (EEG), and magnetic resonance imaging (MRI) to understand the neural oscillatory basis of output-gating. The first session of the experiment will be screening session, in which participants provide written consent to participate, screened for colorblindness, complete questionnaires, and perform a working memory task with retrospective cues. Participants will be invited back to the second session if they show a benefit to their working memory percent correct by use of the informative retro-cue relative to the uninformative neutral cue. This session will also be used to select the number of items that will be used in the working memory task for subsequent sessions. The criteria for difficulty titration is task performance between 60% and 85% correct for retro-cue trials and a benefit of at least 5% greater than neutral cue trials. Thus, different participants will perform the task with different numbers of items to be encoded into working memory. Titration of task difficulty as described here is critical for experiments that use causal manipulation (e.g. transcranial magnetic stimulation) to modulate performance. If participants are performing at ceiling (close to 100%) or at floor (close to random change), then any experimental manipulation of behavior is less likely to impact performance as the task is too "easy" or too "hard." For the second session of the experiment, participants perform the working memory retro-cue task while EEG is recorded. In addition, participants will complete a simple perception color task in which participants see a color and choose the matching color from the color circle. This task tests for the precision of perception throughout the color circle. The EEG data from the second session will be preprocessed and a Morlet wavelet convolution analysis will be conducted. The resulting spectrogram will be contrasted between the informative retro-cue and uninformative neutral cue to derive the theta frequency with peak amplitude in prefrontal cortex, and contrasted between a leftward and rightward retro-cue to derive the alpha frequency with peak amplitude in parietal cortex. These peak frequencies will be used for stimulation in the fourth and fifth session. In the third session, the investigators will acquire structural and functional MRI for each participant. The functional MRI data will be analyzed to identify regions in the anterior middle frontal gyrus and posterior intraparietal sulcus that are functionally connected within the frontal-parietal, "executive control," network. A previous meta-analysis of functional MRI studies found that the regions with peak retro-cue activity was at Montreal Neurological Institute coordinates (-40, 36, 28) for anterior middle frontal gyrus and (-38, -48, 44) for inferior intraparietal sulcus. Therefore, the investigators will constrain the search light to the anatomical landmarks and these coordinates. The center of mass in these regions will be used for targeting with TMS in the subsequent fourth and fifth sessions. In the fourth and fifth sessions, stimulation will be delivered at the timing relative to retro-cue, frequency, and spatial location based on previous localizers. During stimulation, the location of the TMS coil needs to be aligned to the targeted brain region with neuro-navigation software that records the accuracy of each TMS pulse relative to the target. On each trial, the stimulation type will be randomly selected, counter-balanced, and inter-mixed. The effects of rhythmic TMS are not expected to last for more than a few cycles beyond stimulation itself. Therefore, the experimental design randomly intermixes the stimulation type within every task block.

The study 'Theta Connectivity in Working Memory (STAR)', NCT05204381, investigated alpha and theta frequency neural oscillations in the context of cognitive control. Following study completion and during data analysis, a previously unrecognized error in the code of the randomization software used in the conduct of the trial was identified. As a function of the software error, group allocation did not occur as intended and the study design became, de facto and post hoc, a parallel arm design with participants receiving either alpha stimulation or theta stimulation in both stimulation sessions, as opposed to alpha stimulation then theta stimulation in a counterbalanced fashion. The outcomes reported herein of the resulting parallel arm design remain a scientifically valid and appropriate design to investigate the roles of alpha and theta oscillations in the context of cognitive control and additionally resulted in greater statistical power to detect a potential difference between groups.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 35
* Right-handed
* Able to provide informed consent
* Have normal to corrected vision without color blindness
* Willing to comply with all study procedures and be available for the duration of the study Speak and understand English
* Participants will be invited back to the second session only if they are able to perform the task. The criteria for demonstrating the cognitive process of interest is that participants must show a benefit to their working memory percent correct during trials with an informative retro-cue relative to trials with an uninformative neutral cue

Exclusion Criteria:

* Attention Deficit Hyperactivity Disorder (ADHD) (currently under treatment)
* Neurological disorders and conditions, including, but not limited to:
* History of epilepsy
* Seizures (except childhood febrile seizures) Dementia
* History of stroke
* Parkinson's disease
* Multiple sclerosis
* Cerebral aneurysm
* Brain tumors
* Medical or neurological illness or treatment for a medical disorder that could interfere with study participation (e.g., unstable cardiac disease, HIV/AIDS, malignancy, liver or renal impairment)
* Prior brain surgery
* Any brain devices/implants, including cochlear implants and aneurysm clips
* History of current traumatic brain injury
* Failure to pass a colorblindness test
* (For females) Pregnancy or breast feeding
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From 9 to 36 months following publication
Access Criteria: Investigator who proposes to use the data has IRB, IEC, or REB approval and an executed data use/sharing agreement with the University of North Carolina at Chapel Hill.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sessions prior to randomization: Session 1 (S1;baseline behavioral task), Session 2 (S2;baseline EEG), Session 3 (S3;MRI). 71 participants enrolled in S1 (n=1 did not complete, n=13 excluded for performance). n=7 lost to follow-up prior to S2. 50 started S2 (n=1 excluded for performance). n=3 lost to follow-up prior to S3. 46 participants started S3 (n=1 excluded, MRI contraindication). n=6 lost to follow-up prior to S4. 39 participants were randomized to intervention groups.
Groups:
- Theta Stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to frontal and parietal cortex during performance of a cognitive control task while electroencephalography (EEG) is recorded. In the 4th and 5th sessions, TMS is delivered in near-zero phase lag theta-frequency, anti-synchrony theta-frequency, near-zero phase lag arrhythmic-in-synchrony, and arrhythmic-independent TMS. The near-zero phase lag arrhythmic-in-synchrony and arrhythmic-independent TMS is delivered in both the 4th and 5th session to serve as an active control.
  Theta-frequency near-zero phase lag stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in theta-frequency (approximately 6 Hz) with a near-zero phase lag.
  Theta-frequency anti-synchrony stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in theta-frequency (approximately 6 Hz) with a 180 degree phase offset, anti-synchrony.
  Arrhythmic near-zero phase lag stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in an arrhythmic pattern with a near-zero phase lag matched in duration to the rhythmic stimulation for that session.
  Arrhythmic independent stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in different independent arrhythmic patterns matched in duration to the rhythmic stimulation for that session.
- Alpha Stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to frontal and parietal cortex during performance of a cognitive control task while electroencephalography (EEG) is recorded. In the 4th and 5th sessions, TMS is delivered in near-zero phase lag alpha-frequency, anti-synchrony alpha-frequency, near-zero phase lag arrhythmic-in-synchrony and arrhythmic-independent TMS. The near-zero phase lag arrhythmic-in-synchrony and arrhythmic-independent TMS is delivered in both the 4th and 5th session to serve as an active control.
  Arrhythmic near-zero phase lag stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in an arrhythmic pattern with a near-zero phase lag matched in duration to the rhythmic stimulation for that session.
  Arrhythmic independent stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in different independent arrhythmic patterns matched in duration to the rhythmic stimulation for that session.
  Alpha-frequency near-zero phase lag stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in alpha-frequency (approximately 10 Hz) with a near-zero phase lag.
  Alpha-frequency anti-synchrony stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in alpha-frequency (approximately 10 Hz) with a 180 degree phase offset, anti-synchrony.
Period: Session 4
Arm/Group | Theta Stimulation | Alpha Stimulation
Started | 16 | 23
Completed | 15 | 21
Not Completed | 1 | 2
Period: Washout (At Least 1 Day)
Arm/Group | Theta Stimulation | Alpha Stimulation
Started | 15 | 21
Completed | 15 | 18
Not Completed | 0 | 3
Period: Session 5
Arm/Group | Theta Stimulation | Alpha Stimulation
Started | 15 | 18
Completed | 15 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Theta Stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to frontal and parietal cortex during performance of a cognitive control task while electroencephalography (EEG) is recorded. In the 4th and 5th sessions, TMS is delivered in near-zero phase lag theta-frequency, anti-synchrony theta-frequency, near-zero phase lag arrhythmic-in-synchrony, and arrhythmic-independent TMS. The near-zero phase lag arrhythmic-in-synchrony and arrhythmic-independent TMS is delivered in both the 4th and 5th session to serve as an active control.
- Alpha Stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to frontal and parietal cortex during performance of a cognitive control task while electroencephalography (EEG) is recorded. In the 4th and 5th sessions, TMS is delivered in near-zero phase lag alpha-frequency, anti-synchrony alpha-frequency, near-zero phase lag arrhythmic-in-synchrony and arrhythmic-independent TMS. The near-zero phase lag arrhythmic-in-synchrony and arrhythmic-independent TMS is delivered in both the 4th and 5th session to serve as an active control.
- Total: Total of all reporting groups
Arm/Group | Theta Stimulation | Alpha Stimulation | Total
Number analyzed (Participants) | 16 | 23 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 23 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.4 (4.0) | 22.0 (3.7) | 21.7 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 5 | 9 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 16 | 19 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 15 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 23 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Remembered Items
Description: The number of remembered items, often referred to as working memory capacity, is calculated as the number of items to be remembered (2, 3, or 4) times the hit rate minus the false alarm rate, divided by one minus the false alarm rate. The range of values is 0 to 4 where larger values mean better performance.
Time Frame: Measured concurrent with stimulation throughout a 3-hour session
Population: Arrhythmic near-zero phase lag stimulation and Arrhythmic independent stimulation were delivered in both intervention arms (Theta stimulation arm AND Alpha stimulation arm); therefore, the number analyzed for Arrhythmic near-zero phase lag stimulation and Arrhythmic independent stimulation includes all randomized participants from both arms.
Measure: Mean (Standard Deviation); unit: remembered items
Groups:
- Theta-frequency Near-zero Phase Lag Stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in theta-frequency (approximately 6 Hz) with a near-zero phase lag.
  This intervention was only delivered in the Theta stimulation arm.
- Theta-frequency Anti-synchrony Stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in theta-frequency (approximately 6 Hz) with a 180 degree phase offset, anti-synchrony.
  This intervention was only delivered in the Theta stimulation arm.
- Arrhythmic Near-zero Phase Lag Stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in an arrhythmic pattern with a near-zero phase lag matched in duration to the rhythmic stimulation for that session.
  This active control stimulation was delivered in both arms of the study (Theta stimulation intervention arm AND Alpha stimulation intervention arm).
- Arrhythmic Independent Stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in different independent arrhythmic patterns matched in duration to the rhythmic stimulation for that session.
  This active control stimulation was delivered in both arms of the study (Theta stimulation intervention arm AND Alpha stimulation intervention arm).
- Alpha-frequency Near-zero Phase Lag Stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in alpha-frequency (approximately 10 Hz) with a near-zero phase lag.
  This intervention was only delivered in the Alpha stimulation arm.
- Alpha-frequency Anti-synchrony Stimulation: Rhythmic transcranial magnetic stimulation (TMS) is delivered to both frontal and parietal cortex in alpha-frequency (approximately 10 Hz) with a 180 degree phase offset, anti-synchrony.
  This intervention was only delivered in the Alpha stimulation arm.
Arm/Group | Theta-frequency Near-zero Phase Lag Stimulation | Theta-frequency Anti-synchrony Stimulation | Arrhythmic Near-zero Phase Lag Stimulation | Arrhythmic Independent Stimulation | Alpha-frequency Near-zero Phase Lag Stimulation | Alpha-frequency Anti-synchrony Stimulation
Number analyzed (Participants) | 15 | 15 | 33 | 33 | 18 | 18
remembered items | 1.72 (0.48) | 1.68 (0.42) | 1.68 (0.38) | 1.65 (0.37) | 1.71 (0.38) | 1.72 (0.40)
Statistical Analysis 1: Comparison: Theta-frequency Near-zero Phase Lag Stimulation vs Theta-frequency Anti-synchrony Stimulation vs Arrhythmic Near-zero Phase Lag Stimulation vs Arrhythmic Independent Stimulation vs Alpha-frequency Near-zero Phase Lag Stimulation vs Alpha-frequency Anti-synchrony Stimulation; Mixed-factors ANOVA for the interaction between stimulation frequency (theta or alpha) and synchrony (in-phase or anti-phase); Test type: Other; p = 0.783, ANOVA; F-statistic is 0.077

2. Primary Outcome: Strength of Functional Connectivity Between Frontal and Parietal Cortex in Theta-frequency
Description: Functional connectivity will be measured using weighted phase lag index (wPLI) which is the mean of the imaginary component of the difference in theta-frequency phase between frontal and parietal electrical activity during the second half of the stimulation train for every trial. The values range from 0 to 1 where a greater value represents greater functional connectivity.
Time Frame: Measured concurrent with stimulation throughout a 3-hour session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: weighted phase lag index
Arm/Group | Theta-frequency Near-zero Phase Lag Stimulation | Theta-frequency Anti-synchrony Stimulation | Arrhythmic Near-zero Phase Lag Stimulation | Arrhythmic Independent Stimulation | Alpha-frequency Near-zero Phase Lag Stimulation | Alpha-frequency Anti-synchrony Stimulation
Number analyzed (Participants) | 15 | 15 | 33 | 33 | 18 | 18
weighted phase lag index | 0.143 (0.118) | 0.167 (0.158) | 0.116 (0.074) | 0.086 (0.057) | 0.149 (0.104) | 0.156 (0.126)
Statistical Analysis 1: Comparison: Theta-frequency Near-zero Phase Lag Stimulation vs Theta-frequency Anti-synchrony Stimulation vs Arrhythmic Near-zero Phase Lag Stimulation vs Arrhythmic Independent Stimulation vs Alpha-frequency Near-zero Phase Lag Stimulation vs Alpha-frequency Anti-synchrony Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.965, ANOVA; F-statistic is 0.002

3. Secondary Outcome: Average Phase Lag of Functional Connectivity Between Frontal and Parietal Cortex in Theta-frequency
Description: Phase lag is calculated as the resulting phase angle after averaging the phase difference between frontal and parietal cortex electrical signals during the second half of the stimulation train for every trial. The values range from 0 to 360 degrees. A value closer to 0 degrees or closer to 360 degrees represent a near-zero phase lag, where as a value closer to 180 degree represent a larger phase lag.
Time Frame: Measured concurrent with stimulation throughout a 3-hour session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Theta-frequency Near-zero Phase Lag Stimulation | Theta-frequency Anti-synchrony Stimulation | Arrhythmic Near-zero Phase Lag Stimulation | Arrhythmic Independent Stimulation | Alpha-frequency Near-zero Phase Lag Stimulation | Alpha-frequency Anti-synchrony Stimulation
Number analyzed (Participants) | 15 | 15 | 33 | 33 | 18 | 18
degrees | 182.2 (5.73) | 177.4 (14.43) | 182.2 (4.16) | 181.2 (4.32) | 183.1 (6.03) | 183.1 (6.69)
Statistical Analysis 1: Comparison: Theta-frequency Near-zero Phase Lag Stimulation vs Theta-frequency Anti-synchrony Stimulation vs Arrhythmic Near-zero Phase Lag Stimulation vs Arrhythmic Independent Stimulation vs Alpha-frequency Near-zero Phase Lag Stimulation vs Alpha-frequency Anti-synchrony Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.089, ANOVA; F-statistic is 3.046

ADVERSE EVENTS:
Time Frame: Adverse Events were not assessed prior to randomization and group assignment at the start of Session 4. Adverse Events were monitored at Session 4 (up to 3 hours) and Session 5 (up to 3 hours). A systematic assessment was conducted at the end of Session 4 and at the end of Session 5.
Description: A stimulation adverse effects questionnaire was used based on common side effects experience with TMS. This questionnaire was administered at the end of each session in which the participant receives TMS (sessions 4 and 5). This questionnaire was used as a safety measure and to collect data on participant experience. Following the questionnaire, a structured interview was conducted as needed based upon responses on the stimulation adverse effects questionnaire.
Arm/Group | Theta Stimulation | Alpha Stimulation
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/23
Other Adverse Events (participants affected / at risk) | 2/16 | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Theta Stimulation (N=16) | Alpha Stimulation (N=23)
Trouble concentrating (General disorders) | 1 (1) | 1 (1)
Scalp pain (General disorders) | 0 (0) | 1 (1)
Change in Mood (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT05204381/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT05204381/ICF_000.pdf